CLINICAL TRIAL: NCT04720794
Title: A Study To Evaluate The Performance of the Lucira Health All-In-One COVID-19 Test Kit As Compared To The Hologic Panther Fusion SARS-CoV-2 RT-PCR Assay
Brief Title: A Study To Evaluate The Performance of the Lucira Health All-In-One COVID-19 Test Kit vs Hologic Panther Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucira Health Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07A-CLI-006
Record Dates: First submitted 2020-10-13; First posted 2021-01-22 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Covid19; SARS (Severe Acute Respiratory Syndrome); Corona Virus Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Subject Self-Collection and Specimen Testing (Other): Subjects will be provided with the Lucira COVID-19 Test Kit and collect one (1) nasal swab according to the QRI and test the sample on the Lucira COVID-19 All-In-One Test. HCP will observe subject during this process and document any observations and deviations from the QRI.
  Interventions: Device: Lucira COVID-19 All-In-One test kit

INTERVENTIONS:
Device: Lucira COVID-19 All-In-One test kit — The Lucira COVID-19 All-In-One Test Kit is intended to detect the novel coronavirus SARS-CoV-2 that causes COVID-19 in nasal swab samples. This test is a single-use test kit that determines whether there is active shedding of the virus which causes COVID-19. This test utilizes a molecular amplification technology for the detection of SARS-CoV-2 RNA.
  Positive results are indicative of active infection with SARS-CoV-2. Persons who test positive should self-isolate and seek care from their healthcare provider.
  Negative results do not preclude SARS-CoV-2 infection. Persons who continue to experience COVID-like symptoms should seek follow up care from their healthcare provider

SUMMARY:
This Lucira COVID-19 All-In-One Test Kit performance study will be used to establish the performance of the Lucira COVID-19 All-In-One Test Kit as compared to a known high sensitivity RT-PCR molecular assay. The results of this study will be used to demonstrate the Lucira COVID-19 'swab to result in 30 minutes' test kit is similar in performance to known high sensitivity best-in-class molecular assays performed in high complexity labs.

The results of this study will be combined with other studies the Sponsor has underway and will support a FDA Emergency Use Authorization (EUA) of the Lucira COVID-19 All-In-One Test Kit.

This performance study will include nasal swabs self-collected by study subjects at community-based locations with trained medical staff.

A subject's participation in this study will consist of one study visit and one collection event. The subject self-collects a nasal swab sample according to Lucira COVID-19 Test Kit instructions and runs test according to Quick Reference Instructions (QRI).

Following the Lucira COVID-19 All-In-One Test Kit self-collection will be an additional swab collection for reference method testing. One (1) additional NS specimen will be collected either by the health care professional or self-collection, prepared in Transport Medium and sent to a reference laboratory.

DETAILED DESCRIPTION:
The study is a prospective, single site study with community-based sampling in high COVID-19 prevalence communities in California. The Investigational device will be tested on-site and the reference samples will be sent to one (1) reference laboratory in the U.S. Testing in the reference laboratory will be performed by trained laboratory personnel. This study, to be performed with medical staff on site, and will include nasal swabs self-collected by study subjects per the QRI.

Community based sampling will be conducted only by trained medical study staff. Study staff will bring all study materials-the Lucira investigational device as well as the reference swab collection kit-to all subjects enrolled in the study. This mobile, outdoor, community-based sampling method will ensure that COVID-symptomatic persons with fever do not travel from their homes, thus risking exposure to others. All medical staff participating in the study will be under the oversight of the study Principal Investigators and wear appropriate PPE during community visits.

A qualified research person will be designated as the Investigator at each site, with the responsibility for oversight of the study in accordance with Good Clinical Practice (GCP) and regulatory requirements. The protocol and subject informed consent will be reviewed by an Institutional Review Board (IRB) and written IRB approval will be issued prior to enrollment of subjects into the study at that site.

A subject's participation in this study will consist of a single visit. Following completion of the informed consent process and a review of Inclusion/Exclusion criteria to determine eligibility, each subject will receive a unique study identification number. Subject demographics including age, sex, race, and ethnicity, will also be collected at this time.

All subjects will be observed during the swabbing collection by the HCP and HCP will document collection details and any collection issues. The HCP will confirm the Lucira COVID-19 Test Kit is running and will interpret the test results once completed. Nasal swabs obtained from self-collection will be discarded after it has been used for testing.

Following the Lucira COVID-19 Test Kit collection will be a collection for reference method testing. A reference swab should not be collected until the Lucira Test Kit is running. The nasal swab reference swab shall be collected in the same manner as the initial collection, prepared in Transport Medium and sent to the Sutter Shared Laboratory.

To evaluate performance, all reference samples collected will be tested using EUA-cleared molecular method:

• Hologic Panther Fusion SARS-CoV-2 RT-PCR Assay *

Reference testing will characterize specimens as negative or positive for SARS-CoV-2. Therefore, sensitivity and specificity of the Lucira COVID-19 Test will be calculated by comparison with the reference methods.

Additional testing on remaining remnant aliquots may be performed to investigate any discrepant and discordant results as needed, and samples may undergo additional testing by other EUA-cleared molecular methods. The Roche Cobas 6800 SARS-CoV-2 assay will be used for discrepant testing.

If subject consents to storage and future testing of samples, any extra remnants at the end of the study will be returned to the Sponsor for storage.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-75
2. Must be able to read and write in English or Spanish
3. Must be willing to try rapid COVID-19 test and self-collect a nasal swab sample in both nostrils
4. Must be one of the following:

   * Currently experiencing a Fever of 100﮲ Fahrenheit and above or self-reports having fever within the past 48 hours, and experiencing at least one (1) additional associated CDC COVID-19 symptom:

     * Cough
     * Shortness of breath or difficulty breathing
     * Fatigue
     * Muscle or body aches
     * Headache
     * New loss of taste or smell
     * Sore throat
     * Congestion or runny nose
     * Nausea or vomiting
     * Diarrhea
   * Previously tested positive for COVID-19 in past 14 days, and experiencing at least one (1) additional associated CDC COVID-19 symptom
   * Currently experiencing at least three (3) additional associated CDC COVID-19 symptoms so long as at least at least one (1) symptom is either: cough, shortness of breath, and/or new loss of taste or smell.

Exclusion Criteria:

1. Currently suffering from nasal trauma such as a nosebleed
2. Received a nasal rinse/wash/aspirates for standard of care testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
COVID-19 Prevalence Rate / Expected Values counts | 3 months
  Study prevalence of SARS-CoV-2 will be summarized by counts and grouped by age
COVID-19 Prevalence Rate / Expected Values percentages | 3 Months
  Study prevalence of SARS-CoV-2 will be summarized by percentages and grouped by age

SECONDARY OUTCOMES:
Collection Performance/ Incidence Rate counts | 3 Months
  Study observations will be summarized by counts:
  * Self-Collection, Self-tested
  * User Experience
Collection Performance/ Incidence Rate percentages | 3 Months
  Study observations will be summarized by percentages:
  * Self-Collection, Self-tested
  * User Experience
Sensitivity and specificity | 3 Months
  Sensitivity and specificity along with their associated 2-sided Wilson Score 95% Confidence Intervals will be estimated for SARS-CoV-2, on the Lucira COVID-19 All-In-One Test in comparison to the reference test

OTHER OUTCOMES:
Invalid Rate | 3 Months
  The invalid rates, along with their associated 2-sided Wilson Score 95% Confidence Intervals will be estimated for SARS-CoV-2 on the Lucira COVID-19 All-In-One Test

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Kochhar, MD, Principal Investigator — Neeraj Kochhar Family Medicine
Locations (1):
- Neeraj Kochhar Family Medicine, Los Gatos, California, United States

IPD SHARING:
Plan to Share IPD: No